CLINICAL TRIAL: NCT03270683
Title: Doppler Sonography of Cerebral Blood Flow for Early Prognostication After Out-of-hospital Cardiac Arrest: the DOTAC Study
Brief Title: Doppler Sonography of Cerebral Blood Flow for Early Prognostication After Out-of-hospital Cardiac Arrest
Acronym: DOTAC
Status: Completed | Type: Observational
Sponsor: Rennes University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 35RC16_3047_DOTAC
Record Dates: First submitted 2017-08-29; First posted 2017-09-01 (Actual); Last update posted 2019-12-27 (Actual); Status verified 2019-12

CONDITIONS: Cardiac Arrest
Keywords: Out-of-hospital cardiac arrest; transcranial Doppler sonography; cerebrovascular circulation; prognosis
MeSH Terms: conditions — Heart Arrest; Out-of-Hospital Cardiac Arrest

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Objective: To assess neurologic prognostication by early Transcranial Doppler Sonography (TCD) in comatose survivors after cardiac arrest.

Design: Prospective study between May 2016 and November 2017 in a medical intensive care unit and cardiac intensive care unit in a university hospital.

Patients: all comatose patients older than 18 years successfully resuscitated from an out-of-hospital cardiac arrest (OHCA). Patients for whom OHCA is associated with traumatic brain injury, no window for TCD measurements, or dead before neurological prognostication are excluded.

DETAILED DESCRIPTION:
The investigators measure the pulsatility index (PI) and diastolic flow velocity (DFV) of the right and left middle cerebral artery during the first 12 h after return of spontaneous circulation (ROSC). The highest value of DFV and the lowest of PI will use for the statistical analysis. Cerebral Performance Category evaluate neurologic outcome at hospital discharge.

Data provided by early TCD after ROSC are associated with neurological outcome. The use of these data could lead to the development of therapeutics improving cerebral perfusion in patient resuscitated from an OHCA.

ELIGIBILITY:
Inclusion Criteria:

* older 18 years
* out-of-hospital cardiac arrest with recovery of spontaneous cardiac activity

Exclusion Criteria:

* transcranial doppler not done or not interpretable
* associated cranial trauma
* died without neurological assessment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients resuscitated from out-of-hospital cardiac arrest
Sampling Method: Non-Probability Sample
Enrollment: 52 (Actual)
Dates: Start 2016-05-02 (Actual); Primary Completion 2017-10 (Actual); Study Completion 2017-10 (Actual)

PRIMARY OUTCOMES:
Evaluate the relation between TCD measurements and neurologic outcome at hospital discharge | 6 months
  Good score = CPC 1-2 and bad score = CPC 3-5

SECONDARY OUTCOMES:
Measurement of pulsatility index | 12 hours
  Evaluate the association between pulsatility index and period of cardiac arrest
Entry of doppler parameters | 6 months
  Identify a doppler parameter than can improve the neurological outcome

CONTACTS AND LOCATIONS:
Overall Officials: Adel Maamar, Dr, Principal Investigator — CHU Rennes
Locations (1):
- CHU Rennes, Rennes, France